CLINICAL TRIAL: NCT04334018
Title: Observational, Multicentre, Investigator and Patient Blinded, Prospective, Randomized Comparator Study of Cardiac Resynchronization Therapy (CRT) Multi Point Pacing (MPP) Compared to Conventional CRT Pacing Response in Heart Failure Patients.
Brief Title: Multi Point Pacing vs. Conventional STUDY PROTOCOL
Acronym: CRT-MPP
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Other studies on the same theme
Sponsor: CMC Ambroise Paré (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: 2017/02
Record Dates: First submitted 2018-01-31; First posted 2020-04-03 (Actual); Last update posted 2020-04-03 (Actual); Status verified 2020-04

CONDITIONS: Compare Two Programming Modalities for CRT Devices in Heart Failure Patients With an Indication for Cardiac Resynchronization Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- conventional CRT (Placebo Comparator)
  Interventions: Device: conventional CRT
- MPP CRT (Experimental)
  Interventions: Device: MPP CRT

INTERVENTIONS:
Device: conventional CRT — Conventional CRT or biventricular pacing "resynchronizes" left ventricular contraction by pacing the right and left ventricles (LV) simultaneously
  Arms: conventional CRT
Device: MPP CRT — CRT with Multipoint pacing (MPP) where pacing can occur from more than one LV site simultaneously
  Arms: MPP CRT

SUMMARY:
The Purpose of this study is to compare two programming modalities for CRT devices in Heart Failure patients with an indication for Cardiac Resynchronization Therapy

ELIGIBILITY:
Inclusion Criteria:

* Patients with indication for CRT (-P or -D) as per ESC guidelines. Ability to provide written informed consent. Optimal Medical Therapy for at least 3 months

Exclusion Criteria:

* < 18 years and younger
* Pregnant or breastfeeding patients
* Non-LBBB patients (RBBB, intra-ventricular delay)
* Non-ambulatory NYHA class IV effort tolerance
* Myocardial infarction within 40 days before enrolment
* Cardiac surgery or revascularization procedure within 3 months before enrolment, or scheduled in the following 6 months
* Atrial Fibrillation (AF) patients unless AV node ablation is performed, or complete AV block is present (to ensure optimal CRT delivery)
* Patients with life expectancy of less than 12 months due to other medical conditions
* Patients who are involved in another investigational study (device or medical)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-03-01 (Estimated); Primary Completion 2023-03-01 (Estimated); Study Completion 2023-03-01 (Estimated)

PRIMARY OUTCOMES:
Outcome 1 | 12 months
  To evaluate the clinical improvement of CRT MPP as compared to conventional CRT in Heart Failure patients with indication for CRT using automated intra-cardiac EGMs analysis (QuickOpt™) for device optimization, in a large multicentre international study.

CONTACTS AND LOCATIONS:
Locations (6):
- France (5):
  - PHc hôpital d'Antibes la Fontonne, Antibes
  - Centre hospitalier de Cannes, Cannes
  - CMC Ambroise Paré, Neuilly-sur-Seine
  - CHU Nice, Nice
  - Centre Hospitalier de Perpignan, Perpignan
- Centre Hospitalier Princesse Grace, Monaco, Monaco

IPD SHARING:
Plan to Share IPD: No